CLINICAL TRIAL: NCT05070572
Title: Measuring Intraabdominal Pressure, Lactic Acid, and Urine Output in Obese Individuals Undergoing Laparoscopic Inguinal Hernia Repair
Brief Title: Measuring Intraabdominal Pressure, Lactic Acid, and Urine Output
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Maimonides Medical Center (Other)
Collaborators: Potrero Medical (Industry)
Responsible Party: Principal Investigator, Christopher Prien, Principal Investigator, Maimonides Medical Center
Other Study IDs: 2021-05-02-MMC
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Intra-Abdominal Hypertension; Inguinal Hernia
MeSH Terms: conditions — Intra-Abdominal Hypertension; Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Accuryn Monitoring System — Utilization of the Accuryn Monitoring System to measure intraabdominal pressure and urine output during laparoscopic inguinal hernia repair surgery.

SUMMARY:
This study serves as a pilot study with the intention to to measure intraabdominal pressure, lactic acid, and urine output in obese individuals undergoing laparoscopic inguinal hernia repair. By measuring these values, the investigators aim to look for correlations between metrics and determine an accurate and precise measurement of IAP during laparoscopic hernia surgery using the Accuryn Monitoring System. By obtaining accurate and precise measurements of IAP during surgery the investigators will be to compare measurements to previous IAP data obtained during daily activities and strenuous movements and any associations with inguinal hernia recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Obese with BMI > 30
* Diagnosis of inguinal hernia
* Qualify for laparoscopic inguinal hernia repair

Exclusion Criteria:

* Previous bowel resections resulting in short bowel
* Extensive abdominal scarring
* BMI < 30
* Fail to qualify for laparoscopic inguinal hernia repair

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be derived from the elective, outpatient surgical practice of the department of general surgery at Maimonides Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Intraabdominal Pressure | 2 hours
  Maximum IAP levels during surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No